CLINICAL TRIAL: NCT01005706
Title: A Pilot Study Comparing Two Different Sirolimus-based Transition Regimens in African-American Renal Transplant Recipients
Brief Title: Sirolimus Conversions in African-American Renal Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Wyeth Study - HR 19042; HR19042
Record Dates: First submitted 2009-10-09; First posted 2009-11-02 (Estimated); Results first posted 2016-03-11 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2014-02

CONDITIONS: Absence; Kidney
MeSH Terms: interventions — Sirolimus; Mycophenolic Acid; Steroids; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tacrolimus Withdrawal Arm (Active Comparator): At the time of transition patients randomized into this arm of the study will receive loading doses of sirolimus for two days and then 5mg PO daily. Twenty-four hour troughs will be checked per the schedule to ensure and monitor the therapeutic concentrations of 8-12ng/ml.
  Patients randomized into this arm of the study will continue their current dosing regimen and frequency of mycophenolate mofetil. Serum trough level monitoring of mycophenolic acid will not be performed unless clinically warranted per standard of care and dosage adjustments from such levels will be made only with consent of the study primary investigator.
  Interventions: Drug: rapamune, mycophenolate mofetil and steroid
- Tacrolimus Minimization Arm (Active Comparator): Tacrolimus dosing is based on 12-hour whole blood trough concentrations. Target blood concentration is 2-5 ng/ml.
  At the time of transition patients randomized into this arm of the study will receive loading doses of Sirolimus for two days and then 5mg PO daily. Twenty-four hour troughs will be checked per the schedule to ensure and monitor the therapeutic concentrations of 8-12ng/ml.
  Interventions: Drug: tacrolimus, sirolimus and steroid

INTERVENTIONS:
Drug: rapamune, mycophenolate mofetil and steroid — At the time of transition patients randomized into this arm of the study will receive loading doses of sirolimus for two days and then 5mg PO daily. Twenty-four hour troughs will be checked per the schedule to ensure and monitor the therapeutic concentrations of 8-12ng/ml.
  Patients randomized into this arm of the study will continue their current dosing regimen and frequency of mycophenolate mofetil. Serum trough level monitoring of mycophenolic acid will not be performed unless clinically warranted per standard of care and dosage adjustments from such levels will be made only with consent of the study primary investigator.
  Other Names: rapamune (Sirolimus); mycophenolate mofetil (Cellcept)
  Arms: Tacrolimus Withdrawal Arm
Drug: tacrolimus, sirolimus and steroid — Tacrolimus dosing is based on 12-hour whole blood trough concentrations. Target blood concentration is 2-5 ng/ml.
  At the time of transition patients randomized into this arm of the study will receive loading doses of Sirolimus for two days and then 5mg PO daily. Twenty-four hour troughs will be checked per the schedule to ensure and monitor the therapeutic concentrations of 8-12ng/ml.
  Other Names: tacrolimus (Prograf); rapamune (Sirolimus)
  Arms: Tacrolimus Minimization Arm

SUMMARY:
This study's focus is to compare the level effectiveness and safety of regimens involving Sirolimus, Cellcept and steroid to Prograf, Sirolimus and steroid in African-American recipients of kidney transplants.

DETAILED DESCRIPTION:
A major concern in transplantation is finding a successful regimen of medications to lower the potential for the body to reject the newly transplanted organ. The regimens in kidney transplantation include tacrolimus, sirolimus, mycophenolate mofetil and steroids. This study will compare the effectiveness and safety of a regimen including Sirolimus, Prograf, and steroids compared to a regimen including Sirolimus, Cellcept and steroids. These regimens have already been researched in the Caucasian population, and both drug regimens are FDA approved. This study's focus is on the effectiveness and safety of these regimens in African-Americans.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and able to give informed consent
* African-American ethnicity
* Received a first or second non-ECD cadaveric or living donor renal transplant
* Transplant occurred during the past 6 to 24 weeks
* Patient has stable graft function, defined as no change of greater than 30% of baseline serum creatinine during the past month and no acute rejection in the past 6 weeks
* Estimated GFR using the modified MDRD equation of at least 40 mL/min10 at time of enrollment into the study
* Currently receiving tacrolimus, mycophenolate mofetil (at least 1 gm per day), and corticosteroids as their immunosuppression regimen.

Exclusion Criteria:

* Biopsy proven acute rejection episode that occurred within the past 6 weeks
* Malignancy within the past 3 years, except for non-melanoma skin cancer
* Any known intolerances to current immunosuppressant regimen necessitating withdrawal of the offending agent
* Currently enrolled in an investigational trial
* Woman of child bearing potential not utilizing an effective form of birth control
* Patients with uncontrolled dyslipidemia, defined at serum fasting LDL >200 mg/dL or serum fasting triglycerides >500 mg/dL.
* Patients with a spot urine protein to creatinine ratio of > 800 mg of protein per gram of creatinine.
* WBC < 3,000 cells/mm3
* Platelets < 100,000 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2013-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bratton, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- The Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Kahan BD, Camardo JS. Rapamycin: clinical results and future opportunities. Transplantation. 2001 Oct 15;72(7):1181-93. doi: 10.1097/00007890-200110150-00001. No abstract available. PMID 11602840
- [Background] Sehgal SN. Rapamune (RAPA, rapamycin, sirolimus): mechanism of action immunosuppressive effect results from blockade of signal transduction and inhibition of cell cycle progression. Clin Biochem. 1998 Jul;31(5):335-40. doi: 10.1016/s0009-9120(98)00045-9. PMID 9721431
- [Background] MacDonald A, Scarola J, Burke JT, Zimmerman JJ. Clinical pharmacokinetics and therapeutic drug monitoring of sirolimus. Clin Ther. 2000;22 Suppl B:B101-121. doi: 10.1016/s0149-2918(00)89027-x. PMID 10823378
- [Background] Ingle GR, Sievers TM, Holt CD. Sirolimus: continuing the evolution of transplant immunosuppression. Ann Pharmacother. 2000 Sep;34(9):1044-55. doi: 10.1345/aph.19380. PMID 10981252
- [Background] El-Sabrout R, Delaney V, Butt F, Qadir M, Hanson P, Tuteja S, McCollum DA, Butt K. Improved freedom from rejection after a loading dose of sirolimus. Transplantation. 2003 Jan 15;75(1):86-90. doi: 10.1097/00007890-200301150-00016. PMID 12544877
- [Background] Podder H, Stepkowski SM, Napoli KL, Clark J, Verani RR, Chou TC, Kahan BD. Pharmacokinetic interactions augment toxicities of sirolimus/cyclosporine combinations. J Am Soc Nephrol. 2001 May;12(5):1059-1071. doi: 10.1681/ASN.V1251059. PMID 11316866
- [Background] Groth CG, Backman L, Morales JM, Calne R, Kreis H, Lang P, Touraine JL, Claesson K, Campistol JM, Durand D, Wramner L, Brattstrom C, Charpentier B. Sirolimus (rapamycin)-based therapy in human renal transplantation: similar efficacy and different toxicity compared with cyclosporine. Sirolimus European Renal Transplant Study Group. Transplantation. 1999 Apr 15;67(7):1036-42. doi: 10.1097/00007890-199904150-00017. PMID 10221490
- [Background] MacDonald A. Improving tolerability of immunosuppressive regimens. Transplantation. 2001 Dec 27;72(12 Suppl):S105-12. PMID 11833142
- [Derived] Fleming JN, Taber DJ, Pilch NA, McGillicuddy JW, Srinivas TR, Baliga PK, Chavin KD, Bratton CF. A randomized, prospective comparison of transition to sirolimus-based CNI-minimization or withdrawal in African American kidney transplant recipients. Clin Transplant. 2016 May;30(5):528-33. doi: 10.1111/ctr.12718. Epub 2016 Mar 14. PMID 26914542

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tacrolimus Withdrawal Arm | Tacrolimus Minimization Arm
Started | 23 | 17
Completed | 23 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tacrolimus Withdrawal Arm | Tacrolimus Minimization Arm | Total
Number analyzed (Participants) | 23 | 17 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (14) | 54 (11) | 52 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 19 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness and Safety of a Particular Drug Regimen to Prevent Kidney Rejection
Description: Number of Participants with Kidney Rejections
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Tacrolimus Withdrawal Arm | Tacrolimus Minimization Arm
Number analyzed (Participants) | 23 | 17
participants | 4 | 1

ADVERSE EVENTS:
Arm/Group | Tacrolimus Withdrawal Arm | Tacrolimus Minimization Arm
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/17
Other Adverse Events (participants affected / at risk) | 11/23 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Withdrawal Arm (N=23) | Tacrolimus Minimization Arm (N=17)
Death (General disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Withdrawal Arm (N=23) | Tacrolimus Minimization Arm (N=17)
Infection (Infections and infestations) | 8 | 11
CMV (Immune system disorders) | 1 | 2
BK Viremia (Immune system disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No